CLINICAL TRIAL: NCT00743093
Title: Aminotransferase Trends During Prolonged Therapeutic Acetaminophen Dosing
Brief Title: Aminotransferase Trends During Prolonged Acetaminophen Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, Kennon Heard, Fellowship Director, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: COMIRB #06-1265
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Drug Toxicity; Healthy
Keywords: acetaminophen; protein adducts; drug safety; alanine aminotransferase; Alanine Amino Transferase
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetaminophen (Experimental): acetaminophen, 4 grams/day (1 gram every 4 hours for 4 doses)
  Interventions: Drug: acetaminophen
- placebo (Placebo Comparator): placebo for acetaminophen 4 grams/day (2 caplets every 4 hours for 4 doses)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acetaminophen — 500 mg caplets; 2 caplets (1 g)/dose; 4 doses (4 g)/day, 4 hours apart for 16 to 40 days.
  Other Names: tylenol
  Arms: acetaminophen
Drug: placebo — placebo caplets, 2 caplets per dose, 4 doses per day, 4 hours apart for 16 to 40 days
  Arms: placebo

SUMMARY:
The objective of this study is to monitor liver function tests (blood levels of an indicator of liver function) of healthy people taking the maximum labeled daily dose of acetaminophen compared to people taking placebo for 16 to 40 days. Those people that continue to have normal liver tests after 16 days will have completed their part of the study. People that develop abnormal liver function tests will continue taking acetaminophen or placebo, and have their liver tests monitored closely for up to an additional 24 days. This is to (1) make sure these tests return to normal and (2) determine when these tests return to normal while still taking acetaminophen or placebo. If at any time the liver tests indicate anything more than a minor increase, you would be immediately told to stop taking the study drug.

Secondary objective is to determine the proportion of subjects that have detectable acetaminophen-protein adducts after daily dosing.

DETAILED DESCRIPTION:
Acetaminophen use is common and many consumers take 4g/day for longer than 4 days. The use of 4g/day of acetaminophen for more than 4 days causes an asymptomatic ALT elevation in some people. This elevation most likely resolves while continuing treatment, but it is possible that some individuals may go on to develop clinical liver injury. By carefully following healthy subjects who are taking the maximal daily dose of acetaminophen, we can safely determine if the ALT elevation resolves or progresses to clinical liver injury. If a subject develops clinical liver injury we can intervene before irreversible injury occurs.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older

Exclusion Criteria:

1. History of acetaminophen ingestion on any of the four days preceding study enrollment
2. Measurable serum acetaminophen level at time of enrollment
3. Viral markers of Hepatitis B or C, or viral markers of Hepatitis A with an ALT level greater than ULN during screening laboratory testing
4. Serum ALT or AST level greater than ULN at Screening or Day 0
5. Total bilirubin level greater than ULN at Screening or Day 0
6. INR level greater than ULN at Screening
7. Alkaline phosphatase level greater than ULN at Screening
8. Platelet count less than 125 10^9/L at Screening
9. Known cholelithiasis
10. Positive pregnancy test at Screening (female participants only)
11. History of consuming more than an average of 3 alcohol containing drinks daily over the preceding 2 weeks
12. History of consuming 3 or more alcohol containing drinks on any given day during the 2 weeks prior to study enrollment
13. New prescription medication started within the previous 30 days
14. Currently taking isoniazid
15. Currently taking warfarin
16. Currently adheres to a fasting type diet as determined by self report
17. Currently has anorexia nervosa as determined by self report
18. Participant is clinically intoxicated, psychiatrically impaired or unable to give informed consent for any reason
19. Known hypersensitivity or allergy to acetaminophen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kennon Heard, MD, Principal Investigator — Denver Health/Rocky Mountain Poison & Drug Center
Locations (2):
- United States (2):
  - University of Colorado Health Sciences Center - GCRC, Aurora, Colorado
  - Denver Health Rocky Mountain Poison and Drug Center, Denver, Colorado

REFERENCES:
- [Background] Drug Induced Liver Injury Network, U. S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER). Guidance for Industry Drug Induced Liver Injury: Premarketing Clinical Evaluation [Web Page]. 2007 Oct; Accessed 2008 Jan 17. Available at: http://www.fda.gov/cder/guidance/index.htm.
- [Background] Case JP, Baliunas AJ, Block JA. Lack of efficacy of acetaminophen in treating symptomatic knee osteoarthritis: a randomized, double-blind, placebo-controlled comparison trial with diclofenac sodium. Arch Intern Med. 2003 Jan 27;163(2):169-78. doi: 10.1001/archinte.163.2.169. PMID 12546607
- [Background] Davern TJ 2nd, James LP, Hinson JA, Polson J, Larson AM, Fontana RJ, Lalani E, Munoz S, Shakil AO, Lee WM; Acute Liver Failure Study Group. Measurement of serum acetaminophen-protein adducts in patients with acute liver failure. Gastroenterology. 2006 Mar;130(3):687-94. doi: 10.1053/j.gastro.2006.01.033. PMID 16530510
- [Background] Garcia Rodriguez LA, Gonzalez-Perez A. Long-term use of non-steroidal anti-inflammatory drugs and the risk of myocardial infarction in the general population. BMC Med. 2005 Nov 29;3:17. doi: 10.1186/1741-7015-3-17. PMID 16316472
- [Background] Golden HE, Moskowitz RW, Minic M. Analgesic efficacy and safety of nonprescription doses of naproxen sodium compared with acetaminophen in the treatment of osteoarthritis of the knee. Am J Ther. 2004 Mar-Apr;11(2):85-94. doi: 10.1097/00045391-200403000-00002. PMID 14999359
- [Derived] Heard K, Green JL, Anderson V, Bucher-Bartelson B, Dart RC. A randomized, placebo-controlled trial to determine the course of aminotransferase elevation during prolonged acetaminophen administration. BMC Pharmacol Toxicol. 2014 Jul 22;15:39. doi: 10.1186/2050-6511-15-39. PMID 25047090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from August 2008 through August 2011 in the Denver Metro area. Healthy volunteers were recruited from the community through the use of approved advertisements.
Pre-assignment Details: 398 subjects were consented for the study. Of these, 122 were excluded for not meeting full eligibility criteria. 276 eligible subjects were assigned to treatment groups, of which 252 completed all study requirements.
Groups:
- Acetaminophen Arm: acetaminophen
  acetaminophen : 500 mg caplets; 2 capsules (1 g)/dose; 4 doses (4 g)/day, 4 hours apart for 16 to 40 days.
- Placebo Arm: placebo
  placebo : placebo caplets, 2 caplets per dose, 4 doses per day, 4 hours apart for 16 to 40 days
Period: Base Study Period
Arm/Group | Acetaminophen Arm | Placebo Arm
Started | 224 | 52
Completed | 205 | 47
Not Completed | 19 | 5
Period: Extended Dosing Period
Arm/Group | Acetaminophen Arm | Placebo Arm
Started | 51 (Subjects not meeting stopping criteria after base continued into the extended dosing.) | 1 (Subjects not meeting stopping criteria after base continued into the extended dosing.)
Completed | 48 | 1
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected on all subjects at screening and included: race, ethnicity, gender, age, weight, and height. The number of participants included in the analysis (276) is based on the safety population, which includes any subject that took at least one dose of study medication.
Groups:
- Acetaminophen Arm: acetaminophen 500 mg
- Placebo Arm: placebo
- Total: Total of all reporting groups
Arm/Group | Acetaminophen Arm | Placebo Arm | Total
Number analyzed (Participants) | 224 | 52 | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 221 | 52 | 273
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 36.3 (12.16) | 35.8 (12.50) | 36.2 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 39 | 202
  Male | 61 | 13 | 74
Region of Enrollment [Number; unit: participants]
  United States | 224 | 52 | 276

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Treated With Long-term Acetaminophen (4 g/Day) That Develops Persistent ALT Elevations.
Description: ALT was measured on Day 0 and 16 for all study participants. Subjects with an elevated ALT at Day 16 continued dosing with study drug and continued to have their ALT measured every three days until the ALT elevation resolved or until Day 40. Persistent ALT elevation was defined as any subject with an unresolved ALT elevation at study Day 40.
Time Frame: serial samples for 16-40 days
Population: The total number of subjects completing the trial was used for analysis. Subjects who withdrew early were not included.
Measure: Number; unit: participants
Arm/Group | Acetaminophen Arm | Placebo Arm
Number analyzed (Participants) | 205 | 47
participants
  Subjects without persisitent ALT elevation | 204 | 47
  Subjects with persistent ALT elevation | 1 | 0

2. Secondary Outcome: The Proportion of Subjects With Detectable Serum Acetaminophen-cysteine Adduct (APAP-cys) Concentrations 1, 2, and 3 Days After Starting the Maximal Recommended Dosing of Acetaminophen (4 g/Day).
Time Frame: Days 1-3
Population: A subset of the safety population was monitored for early detection of APAP-cys. This subset of subjects had APAP-cys measured at Days 1, 2, and 3 in addition to other protocol defined timepoints.
Measure: Number; unit: participants
Arm/Group | Acetaminophen Arm | Placebo Arm
Number analyzed (Participants) | 64 | 15
participants
  Day 1-No. Subjects with Detectable APAP-cys | 7 | 1
  Day 2-No. Subjects with Detectable APAP-cys | 57 | 1
  Day 3-No. Subjects with Detectable APAP-cys | 59 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting at the time of consent through study completion.
Arm/Group | Acetaminophen Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/52
Other Adverse Events (participants affected / at risk) | 147/224 | 25/52
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acetaminophen Arm (N=224) | Placebo Arm (N=52)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 | 0
Eye disorders (Eye disorders) | 2 | 0
Gastrointestinal Disorders (Gastrointestinal disorders) | 70 | 10
General disorders and administration site conditions (General disorders) | 23 | 3
Infections and infestations (Infections and infestations) | 14 | 2
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 10 | 2
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 | 1
Muskuloskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 26 | 5
Nervous system disorders (Nervous system disorders) | 42 | 11
Psychiatric disorders (Psychiatric disorders) | 6 | 1
Renal and urinary disorders (Renal and urinary disorders) | 0 | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 5 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 23 | 5
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 9 | 0
Vascular disorders (Vascular disorders) | 9 | 1

LIMITATIONS AND CAVEATS:
This study was limited to healthy volunteers. The ingestion of each dose of study drug and use of other medications was self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No